CLINICAL TRIAL: NCT05107089
Title: Ultrasound Guided Subclavian Vein Cannulation at Emergency Room , Success Rate and Incidence of Complications
Brief Title: Ultrasound Guided Subclavian Vein Cannulation at Emergency Room
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ARMohamed, Resident, Assiut University
Other Study IDs: Subclavian vein cannulation
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Ultrasound Subclavian Cannulation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Use of ultrasound at subclavian vein cannulation for visualization

SUMMARY:
1. To observe and report the success rate associated with the use of ultrasound for subclavian vein catheterization.
2. To observe and report the type and complications and any constrains associated with this technique.

DETAILED DESCRIPTION:
Central venous catheterisation is a commonly performed procedure in anaesthesia, critical care, acute and emergency medicine. 1 , the subclavian vein (SCV) has been an important vessel for central venous cannulation.2 The SCV cannulation offers several advantages when compared to the common alternative sites for central venous access. These advantages may include fewer cases of thrombosis, infectious complications, better patient comfort, and increased ability to remain patent in hypovolemic states.3-4 Traditionally, subclavian venous catheterisation has been performed using the landmark technique and because of the complications associated with this technique, it is not commonly performed.1 the complications such as catheter malposition, arterial puncture, hematoma, pneumothorax, hemothorax, and nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* All patient admitted to emergency room and indicated for central venous catheterization

Exclusion Criteria:

* 1. Any contraindication for central vein cannulation as coagulopathy, hemorrhage from target vessel, suspected proximal vascular injury 2- Age below 18 year

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient has arrived to the emergency room with sign of hypovolemic shock Or arrested
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
success rate of the ultrasound guided subclavian vein cannulation success rate of the ultrasound guided subclavian vein cannulation Success rate of ultrasound guided of subclavian vein cannulation | Baseline
  Use of ultrasound at visualization of cannulation of subclavian vein

REFERENCES:
- [Background] Hayashi M, Oshima K. Purification and properties of oxytocinase (cystine amino-peptidase) from monkey placenta. J Biochem. 1976 Aug;80(2):389-96. doi: 10.1093/oxfordjournals.jbchem.a131288. PMID 12146